CLINICAL TRIAL: NCT04784299
Title: A Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Design Investigation to Evaluate Performance and Safety of YVOIRE Volume Plus Versus Restylane Lyft with Lidocaine for Temporary Improvement of Mid-face Volume
Brief Title: To Evaluate the Performance and Safety of YVOIRE Volume Plus for Improvement of Mid-face Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL029
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Midface Volume Deficit

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YVOIRE volume plus (Experimental): Hyaluronic acid dermal filler
  Interventions: Device: YVOIRE volume plus
- Restylane Lyft with Lidocaine (Active Comparator): Hyaluronic acid dermal filler
  Interventions: Device: Restylane Lyft with Lidocaine

INTERVENTIONS:
Device: YVOIRE volume plus — Hyaluronic acid dermal filler
  Arms: YVOIRE volume plus
Device: Restylane Lyft with Lidocaine — Hyaluronic acid dermal filler
  Arms: Restylane Lyft with Lidocaine

SUMMARY:
A Study to Evaluate the Performance and Safety of YVOIRE volume plus for Temporary Improvement of Mid-face Volume

DETAILED DESCRIPTION:
This is a Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Design Investigation to Evaluate the Performance and Safety of YVOIRE volume plus versus Restylane Lyft with Lidocaine for Temporary Improvement of Mid-face Volume.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged between 21 to 75 years (inclusive)
* 2 or 3 on the 5-point MFVLRS (Mid Face Volume Loss Rating Scale)
* Desire cheek augmentation to correct volume deficit in the midface.
* Agree to use contraception
* Sign Informed Consent Form

Exclusion Criteria:

* have undergone facial plastic surgery, tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent dermal fillers in the midface area
* have undergone temporary facial dermal filler injections with HA-based fillers within 12 months, porcine-based collagen fillers within 24 months prior to screening
* have mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases
* have history of anaphylaxis, multiple severe allergies, or allergy to lidocaine, HA products, or Streptococcal protein
* have history of bleeding disorder
* have a tendency to develop hypertrophic scarring or keloid

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of YVOIRE volume plus versus Restylane Lyft with Lidocaine | 24 weeks from baseline
  To demonstrate non-inferiority of YVOIRE volume plus versus Restylane Lyft with Lidocaine in the improvement of mid face volume by comparing the mean change from Baseline in the Mid Face Volume Loss Rating Scale (MFVLRS) at 24 weeks after the final treatment
Responder rate of YVOIRE volume plus | 24 weeks from baseline
  To confirm performance of YVOIRE volume plus by the responder rate (defined as at least 1-point improvement from Baseline) at 24 weeks after the final treatment

SECONDARY OUTCOMES:
Mean Change of Mid Face Volume Loss Rating Scale (MFVLRS) | 4, 8, 12, 52 weeks from baseline
  To compare the performance of YVOIRE volume plus to Restylane Lyft with Lidocaine based on the MFVLRS
Responder rate of YVOIRE volume plus | 4, 8, 12, 52 weeks from baseline
  To confirm performance of YVOIRE volume plus by the responder rate (defined as at least 1-point improvement from Baseline) at 24 weeks after the final treatment
Mean Score of Mid Face Volume Loss Rating Scale (MFVLRS) | 4, 8, 12, 24, 52 weeks from baseline
  o compare the performance of YVOIRE volume plus to Restylane Lyft with Lidocaine based on the MFVLRS
The mean scores of the GAIS | 4, 8, 12, 24, 52 weeks from baseline
  To compare the performance of YVOIRE volume plus to Restylane Lyft with Lidocaine based on Global Aesthetic Improvement Scale (GAIS)
Mean change in mid-face volume | 24 weeks from baseline
  To compare the performance of YVOIRE volume plus to Restylane Lyft with Lidocaine based on the three dimensional (3-D) photograph measurement

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Principal Investigator — LG Chem Investigational site 01
Locations (1):
- LG Chem investigational site 01, Munich, Germany

IPD SHARING:
Plan to Share IPD: No